CLINICAL TRIAL: NCT01543139
Title: A Double-Blind, Placebo-Controlled Trial of Combined Cytidine- and Creatine-Containing Drug and Dietary Supplement in the Treatment of the Bipolar Depression
Brief Title: Cytidine- and Creatine-Containing Drug in Treating Bipolar Depression
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The research project has been cancelled before any participants were enrolled.
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBI_bipolar2015
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Bipolar Depression
Keywords: Bipolar Depression; Magnetic resonance spectroscopy; Cytidine-; Creatine-
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Valproate+Cytidine-+Creatine- (Experimental): The subjects with bipolar depression, treated with cytidine- and creatine-containing drug and dietary supplement in addition to valproate
  Interventions: Drug: Valproate+Cytidine-+Creatine-
- Valproate+Cytidine- (Active Comparator): The subjects with bipolar depression, treated with cytidine-containing drug and dietary supplement in addition to valproate
  Interventions: Drug: Valproate+Cytidine-
- Valproate (Active Comparator): The subjects with bipolar depression, treated with valproate
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Valproate+Cytidine-+Creatine- — Valproate: Week0-8: 300mg/day, Cytidine-: Week0-8: 2g/day, Creatine-: Week0-1: 3g/day Week1-8: 5g/day
  Arms: Valproate+Cytidine-+Creatine-
Drug: Valproate+Cytidine- — Valproate: Week0-8: 300mg/day, Cytidine-: Week0-8: 2g/day
  Arms: Valproate+Cytidine-
Drug: Valproate — Valproate: Week0-8: 300mg/day
  Arms: Valproate

SUMMARY:
This proposed research is aimed to investigate the efficacy and safety of combined cytidine- and creatine-containing drug and dietary supplement in treating bipolar depression and to evaluate changes in relevant brain biochemical metabolism using magnetic resonance spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* 19-65 year-old male or female
* Bipolar depression diagnosed by Structured Clinical Interview for DSM-IV (SCID-IV)
* Written informed consent

Exclusion Criteria:

* Present use of drugs for bipolar depression or any psychotropic medication
* Use of psychoactive medication that may affect brain imaging findings
* Diagnosis of any other axis I psychiatric disorder
* Presence of borderline personality disorder or antisocial personality disorder
* Presence of any major physical or neurological illness (e.g., epilepsy, multiple sclerosis, brain tumor, cerebrovascular disease, etc.)
* Hypersensitivity to divalproate, valpromide or diagnosis of porphyria
* Past or current liver disease, current severe liver or pancreas dysfunction
* Currently taking mefloquine
* Presence of alcohol or drug dependence, drug abuse
* Intelligence quotient below 80
* Contraindications to magnetic resonance imaging
* Women who are pregnant, breastfeeding, or planning pregnancy
* Allergy or intolerance to the study drugs

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12-01 (Estimated); Primary Completion 2017-04-30 (Estimated); Study Completion 2017-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depressive symptom scores at 4 weeks | Baseline and at 4 weeks
Change from baseline in depressive symptom scores at 8 weeks | Baseline and at 8 weeks

SECONDARY OUTCOMES:
Changes in brain Glx (glutamate+glutamine) level assessed using magnetic resonance spectroscopy at baseline and 8 weeks | Baseline and at 8 weeks
Number of participants with adverse events | 4 weeks
Number of participants with adverse events | 8 weeks
Changes in brain phosphocreatine level assessed using magnetic resonance spectroscopy at baseline and 8 weeks | Baseline and at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: In Kyoon Lyoo, MD, PhD, MMS, Principal Investigator — Ewha Womans University
Locations (1):
- Ewha Womans University Medical Center, Seoul, South Korea